CLINICAL TRIAL: NCT02152891
Title: A Community Paramedicine Initiative for Older Adults Living in Subsidized Housing (CHAP-EMS/Renamed to CP@Clinic)
Brief Title: A Community Paramedicine Initiative for Older Adults Living in Subsidized Housing (CHAP-EMS/CP@Clinic)
Acronym: CHAP-EMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOP-133563
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Diseases; Diabetes Mellitus
Keywords: Emergency Medical Services; Elderly
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHAP-EMS/CP@clinic Program Intervention (Experimental): 12 month implementation of the intervention
  Interventions: Behavioral: CHAP-EMS/CP@clinic
- Control (No Intervention): Will complete a survey at baseline and at 1 year, no program or intervention provided

INTERVENTIONS:
Behavioral: CHAP-EMS/CP@clinic — Community Paramedicine program to assess cardiovascular, diabetes, and fall risk; discuss lifestyle changes and goals; and refer to appropriate resources.
  Arms: CHAP-EMS/CP@clinic Program Intervention

SUMMARY:
Older adults living in subsidized housing report poorer health. Their age and low income make it harder for them to use community services. Many older adults have heart disease and diabetes, which lead to frequent emergency calls and hospital admissions. To decrease the costs of treating heart disease and diabetes through emergency and hospitalization, improved screening and health education is needed. Our program will take place in communal areas within housing buildings of older adults and deliver a heart disease, diabetes, and falls risk check-up with health education. This is expected to improve the health of older adults leading to fewer emergency calls and hospital visits.

ELIGIBILITY:
Inclusion Criteria:

* 55 years and older
* Resides in subsidized apartment building

Exclusion Criteria:

- None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Diabetes Risk (CANRISK) Score | Baseline and 1 year
  The CANRISK tool provides a 10-year risk of diabetes score and will be administered by the paramedic during the CHAP-EMS session.
Change in Blood Pressure | Baseline and after each assessment (up to one year)
  Since the participants are invited to attend the intervention weekly, but are not required to attend, the number of assessments and time of assessments will vary. Multilevel analysis will be conducted that accounts for this variance in repeated measures.
Change in health perceptions, behaviours, and knowledge of resources | Baseline and 1 year
  A face-to-face survey will be administered to determine participant health perceptions, behaviours, and knowledge.
Change in Health Care Utilization | Baseline and 1 year
  Health Care Utilization will be assessed through administrative databases (e.g. hospital visits). Utilization by residents in the intervention apartment buildings will be compared to baseline and compared to the control apartment buildings.
Change in rate of EMS Calls | Baseline and 1 year
  Rate EMS calls by residents in the intervention apartment buildings will be compared to baseline and compared to the control apartment buildings.

CONTACTS AND LOCATIONS:
Overall Officials: Gina Agarawal, Principal Investigator — McMaster University
Locations (5):
- Canada (5):
  - City of Greater Sudbury, Greater Sudbury, Ontario
  - Guelph-Wellington Emergency Medical Services and County of Wellington Social Services Department - Housing Services, Guelph, Ontario
  - Hamilton Paramedic Services, Hamilton, Ontario
  - County of Simcoe, Simcoe, Ontario
  - York Region, York, Ontario

REFERENCES:
- [Derived] Brar J, AlShenaiber L, Dzerounian J, Pirrie M, Angeles R, Marzanek F, Agarwal G. Effects of the Community Paramedicine at Clinic (CP@clinic) program on the health behaviours of older adults residing in social housing: secondary outcomes of a cluster-randomized trial. BMC Public Health. 2025 Mar 6;25(1):887. doi: 10.1186/s12889-025-21997-w. PMID 40050836
- [Derived] Agarwal G, Pirrie M, Angeles R, Marzanek F, Paterson JM, Nguyen F, Thabane L. Community Paramedicine Program in Social Housing and Health Service Utilization: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2441288. doi: 10.1001/jamanetworkopen.2024.41288. PMID 39466243
- [Derived] Marzanek F, Nair K, Ziesmann A, Paramalingam A, Pirrie M, Angeles R, Agarwal G. Perceived value and benefits of the Community Paramedicine at Clinic (CP@clinic) programme: a descriptive qualitative study. BMJ Open. 2023 Nov 21;13(11):e076066. doi: 10.1136/bmjopen-2023-076066. PMID 37989376
- [Derived] Agarwal G, Pirrie M, Angeles R, Marzanek F, Thabane L, O'Reilly D. Cost-effectiveness analysis of a community paramedicine programme for low-income seniors living in subsidised housing: the community paramedicine at clinic programme (CP@clinic). BMJ Open. 2020 Oct 27;10(10):e037386. doi: 10.1136/bmjopen-2020-037386. PMID 33109643
- [Derived] Agarwal G, Angeles R, Pirrie M, McLeod B, Marzanek F, Parascandalo J, Thabane L. Reducing 9-1-1 Emergency Medical Service Calls By Implementing A Community Paramedicine Program For Vulnerable Older Adults In Public Housing In Canada: A Multi-Site Cluster Randomized Controlled Trial. Prehosp Emerg Care. 2019 Sep-Oct;23(5):718-729. doi: 10.1080/10903127.2019.1566421. Epub 2019 Feb 4. PMID 30624150
- [Derived] Agarwal G, Angeles R, Pirrie M, McLeod B, Marzanek F, Parascandalo J, Thabane L. Evaluation of a community paramedicine health promotion and lifestyle risk assessment program for older adults who live in social housing: a cluster randomized trial. CMAJ. 2018 May 28;190(21):E638-E647. doi: 10.1503/cmaj.170740. PMID 29807936
- [Derived] Agarwal G, McDonough B, Angeles R, Pirrie M, Marzanek F, McLeod B, Dolovich L. Rationale and methods of a multicentre randomised controlled trial of the effectiveness of a Community Health Assessment Programme with Emergency Medical Services (CHAP-EMS) implemented on residents aged 55 years and older in subsidised seniors' housing buildings in Ontario, Canada. BMJ Open. 2015 Jun 11;5(6):e008110. doi: 10.1136/bmjopen-2015-008110. PMID 26068514